CLINICAL TRIAL: NCT03107078
Title: Using A Novel Classification System in Intravenous Glucocorticoids Therapy of TAO: A Multi-central, Randomized, Open, Superior Trial
Brief Title: Using A Novel Classification System in Intravenous GCs Therapy of TAO: A Multi-central, Randomized, Open, Superior Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jie Shen (Other Government)
Collaborators: The Fifth Affiliated Hospital of Southern Medical University (Other); Huadu District People's Hospital of Guangzhou (Other); Zhujiang Hospital (Other)
Responsible Party: Sponsor-Investigator, Jie Shen, Vice President;Doctoral Supervisor, The Third Affiliated Hospital of Southern Medical University
Organization: The Third Affiliated Hospital of Southern Medical University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ThirdAffiliatedHospitalOfSMU
Record Dates: First submitted 2017-03-08; First posted 2017-04-11 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Thyroid Associated Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Glucocorticoids; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group Ia (Experimental): I:The increase of fat volume dominates .
  a:The weekly protocol was as follows: 0.5 g glucocorticoids weekly for 6 weeks, followed by 0.25 g weekly for 6 weeks.
  Interventions: Drug: Glucocorticoids
- Group Ib (Experimental): I:The increase of fat volume dominates. b:The "qod" protocol was as follows: 0.5 g glucocorticoids qod. for 3 interval days per month for 3 months.
  Interventions: Drug: Glucocorticoids
- Group IIa (Experimental): II:The increase of extraocular muscles volume dominates .
  a:The weekly protocol was as follows: 0.5 g glucocorticoids weekly for 6 weeks, followed by 0.25 g weekly for 6 weeks.
  Interventions: Drug: Glucocorticoids
- Group IIb (Experimental): II:The increase of extraocular muscles volume dominates . b:The "qod" protocol was as follows: 0.5 g glucocorticoids qod. for 3 interval days per month for 3 months.
  Interventions: Drug: Glucocorticoids

INTERVENTIONS:
Drug: Glucocorticoids — Intravenous Glucocorticoids (GCs)
  Other Names: Methylprednisolone

SUMMARY:
For patients with active moderate-to-severe thyroid associated ophthalmopathy (TAO), the Intravenous Glucocorticoids (GCs) is the recommended therapy. However, the efficacy of GCs is not satisfied. Investigators established a novel classification of TAO for the first time to assess more precisely for better personal treatment.

DETAILED DESCRIPTION:
TAO is one of most common extra thyroid manifestation of dysfunctional thyroid disease. Since the morbidity of TAO has been increasing rapidly, Investigators' team is intended to verify the feasibility of the new type of classification system established by the related parameters of orbital MRI scan. Based on classification, investigators compare the efficacy of two GCs therapy. According to MRI,investigators measure the optimal T2 signal intensity ratio (SIR) for the treatment of TAO, which may help to find a better treatment time for therapy.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnostic standard of TAO is according to Bartley's criteria.
2. Patients with active moderate-to-severe TAO based on 2016 EUGOGO guidelines.
3. CAS≥3/7.
4. None of the patients received any glucocorticoids therapy or orbital radiotherapy in the previous 3 months.

Exclusion Criteria:

1. NOSPECS is 0 or 1.Only signs,no symptoms.Signs include:reduced blink(Stellwag symptoms),two reduced cohesion(Mobius levy),moving slowly on the eyelids(Von Graefe sign),to the point of view,the forehead wrinkled skin should not(Joffroyv levy).
2. Suffering from other eye diseases or wearing contact lenses.
3. Suffering from other autoimmune diseases.
4. Acute and chronic infectious diseases.
5. Diabetic retinopathy or hypertensive fundus lesions.
6. Patients received orbital decompression or other orbital surgery.
7. Suffering from eye trauma or ocular surface disease.
8. Special occupants, and the working environment has obvious air pollution etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients defined as Response for the Glucocorticoids Treatment based on the 7 parameters of eye assessment | 2years
  "Response" was defined as at least three of the following outcome measures:
  1. reduction in lid width by at least 3 mm;
  2. reduction in any of the class 2 NOSPECS signs by at least two grades;
  3. reduction in proptosis by at least 2 mm;
  4. reduction in intraocular pressure by at least 2 mm Hg;
  5. improvement in CAS by at least two points;
  6. improvement in diplopia (disappearance or degrade in degree);
  7. improvement in visual acuity by 1 Snellen line.
Number of patients defined as Deterioration for the Glucocorticoids Treatment based on the 7 parameters of eye assessment | 2years
  "Deterioration" of each parameter was defined as follows:
  1. increase in lid width by at least 3 mm;
  2. increase in any of the class 2 NOSPECS signs by at least two grades;
  3. increase in proptosis by at least 2 mm;
  4. increase in intraocular pressure by at least 2 mm Hg;
  5. increase in CAS by at least two points;
  6. increase in diplopia (new onset or upgrade in degree);
  7. decrease in visual acuity by 1 Snellen line.
Number of patients defined as Unchange for the Glucocorticoids Treatment based on the 7 parameters of eye assessment | 2years
  "Unchanged" was defined as no change or changes smaller than previously defined in any of the mentioned parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- the Third Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Z, Luo Y, Huang Q, Chen Z, Song D, Pan D, Hu S, Jiang W, Cai Q, Feng X, Zhang Q, Weng C, Zhong Q, Zhao T, Li C, Zhang T, Shen J. A Randomized Clinical Trial of Intravenous Methylprednisolone With 2 Protocols in Patients With Graves Orbitopathy. J Clin Endocrinol Metab. 2023 Dec 21;109(1):36-45. doi: 10.1210/clinem/dgad476. PMID 37579198